CLINICAL TRIAL: NCT06839339
Title: A Phase II, Randomized, Positive-controlled, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Single Suprachoroidal Space Injection of AL-001 Ophthalmic Injection in Subjects with Wet Age-related Macular Degeneration (wAMD)
Brief Title: Efficacy and Safety of AL-001 Ophthalmic Injection in Subjects with WAMD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Anlong Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AL-001-02
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Wet Age-related Macular Degeneration (wAMD)
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AL-001 Dose 1 (Experimental): Injection of dose 1
  Interventions: Drug: AL-001
- AL-001 Dose 2 (Experimental): Injection of dose 2
  Interventions: Drug: AL-001
- Aflibercept (Active Comparator): Intravitreal injection
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: AL-001 — Administered via suprachoroidal space injection.
  Arms: AL-001 Dose 1; AL-001 Dose 2
Drug: Aflibercept — Intravitreal injection
  Arms: Aflibercept

SUMMARY:
This Phase II study is designed to evaluate the efficacy and safety of AL-001 ophthalmic injection in patients with wet age-related macular degeneration. Eligible patients, who meet the inclusion/exclusion criteria and have shown an anatomic response to an anti-VEGF (Vascular Endothelial Growth Factor) injection, will be randomized in Cohorts 1 and 2 to receive AL-001 administered via suprachoroidal space injection, Cohort 3 to receive Aflibercept.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 50 and ≤ 85.
2. The study eye was diagnosed with subfoveal active choroidal neovascularization (CNV) lesions secondary to wAMD.
3. The study eye has response to anti-VEGF injections.
4. The subject or their legal representative agrees to participate in this study and signs a written ICF.

Exclusion Criteria:

1. Non-wAMD induced CNV or macular edema in the study eye.
2. Non-wAMD induced eye conditions that may affect central vision or medical history that may seriously affect central vision in the study eye.
3. Uncontrolled glaucoma in the study eye.
4. History of vitreoretinal surgery, antiglaucoma trabeculectomy, or other anti-glaucoma filtering surgery in the study eye.
5. Refractive interstitial opacity that significantly affects visual function assessment or fundus examination in the study eye.
6. Ametropia (high myopia or high hyperopia) > 8.0D in the study eye, or significant posterior scleral staphyloma in the study eye.
7. Malignant tumor in any eye, including but not limited to eye lymphoma or choroidal melanoma.
8. None of intraocular inflammation in the study eye.
9. Other conditions that may affect compliance or may not be suitable to participate in this trial in the opinion of investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of AL-001 on BCVA | Week 24
  Change in BCVA

SECONDARY OUTCOMES:
Safety | Week 56
  Incidence of adverse events (AEs) and serious adverse events (SAEs)
Evaluate the effect of AL-001 on central retinal thickness (CRT) | Week 56
  Mean change from baseline in CRT as measured

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Hospital, Beijing, China